CLINICAL TRIAL: NCT01757938
Title: Shang Ring Versus Forceps-guided Adult Male Circumcision: a Randomized Controlled Effectiveness Study in Southwestern Uganda.
Brief Title: Randomized Control Trial of Shang Ring Versus Forceps-guided Adult Male Circumcision in Southwestern Uganda.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUST2012-1
Record Dates: First submitted 2012-12-19; First posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: HIV
Keywords: HIV; Prevention; Adult Male Circumcision; Uganda; Shang Ring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shang Ring Guided Circumcision (Experimental): The Shang Ring (SR) (Wuhu Santa Medical Devices Technology Co Ltd, China) male circumcision performed by study surgeon (study PI). In both study groups, participants were cleaned with povidone iodine solution and draped in a sterile fashion. Local anesthesia was administered to the dorsal penile nerve and penile ring blocks using 3mg/kg of 1% lidocaine. The surgeon measured participants in the SR group to determine ring size. Patients for whom a suitable ring size was not available crossed over to the FG group, but remained in the SR group for intention to treat (ITT) analyses.
  Interventions: Procedure: Shang Ring Guided Circumcision
- Forceps Guided Circumcision (Active Comparator): Standard forceps guided adult male circumcision was performed. In both study groups, participants were cleaned with povidone iodine solution and draped in a sterile fashion. Local anesthesia was administered to the dorsal penile nerve and penile ring blocks using 3mg/kg of 1% lidocaine.
  Interventions: Procedure: Forceps Guided Circumcision

INTERVENTIONS:
Procedure: Shang Ring Guided Circumcision
  Arms: Shang Ring Guided Circumcision
Procedure: Forceps Guided Circumcision
  Arms: Forceps Guided Circumcision

SUMMARY:
Adult male circumcision (AMC) can reduce the incidence of HIV transmission by 40-60% in sub-Saharan Africa (SSA). The World Health Organisation and Joint United Nations Programme on HIV/AIDS advocate AMC for the reduction of HIV transmission in heterosexual men, and feasibility studies have demonstrated that AMC programmes can be effectively delivered to hyperendemic communities, such as those in SSA. Despite these recommendations, the potential effects of AMC have been attenuated by low uptake, with only 5% of all men who could benefit undergoing surgery to date. Traditional, time-consuming methods of AMC that require formal surgical training limit uptake in low-income countries. Training and implementation by non-physician health providers is dampened by a need to perform approximately 100 procedures to achieve satisfactory operative time and adverse effect rates. The investigators performed a randomised controlled effectiveness study to compare the shang ring (SR) with standard forceps-guided (FG)-AMC in a publicly funded regional referral hospital with a locally trained surgeon in Mbarara, western Uganda.

DETAILED DESCRIPTION:
Male undergoing elective AMC were recruited from the surgical outpatient department of Mbarara Regional Referral Hospital, Uganda. Patient age, marital status, smoking history and motive to seek AMC were recorded for each participant.

The investigators performed block randomization by study day. Consenting participants selected an opaque envelope from a box for randomization to SR or FG groups. All AMC procedures were performed by a locally-trained surgeon who had performed over 100 prior FG procedures but who had no prior experience of the SR procedure.

A study surgeon performed all procedures in the hospital operating theatres. In both study groups, participants were cleaned with povidone iodine solution and draped in a sterile fashion. Local anesthesia was administered to the dorsal penile nerve and penile ring blocks using 3mg/kg of 1% lidocaine. The surgeon measured participants in the SR group to determine ring size. Patients for whom a suitable ring size was not available crossed over to the FG group, but remained in the SR group for intention to treat (ITT) analyses. An assistant measured operative time using a stopwatch. For the SR group, timing began as the ring began to be fitted, and ceased when the foreskin had been excised. For the FG group, timing began at the first incision and ceased when the final suture was completed. Patients were discharged on the day of procedure, provided with sterile gauze dressings, and informed to change them twice daily until the first follow-up appointment.

All pre- and post-operative assessments were performed by the lead investigator at one hour after the procedure, and on the 3rd, 7th, 14th and 21st post-operative days.

The investigators measured incidence rates of all outcomes and estimated relative risk for the SR versus FG groups by fitting Poisson regression models with robust errors. The investigators compared time to healing with Kaplan-Meier survival curves and measured for a difference between groups using the likelihood ratio test. All analyses were initially performed using ITT analysis, and were repeated with an as-treated analysis by reallocating the 7 participants who crossed into the FG group.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Greater than 18 years old
* Desire for adult male circumcision
* Presenting outpatient department of Mbarara Regional Referral Hospital
* Provide written informed consent

Exclusion Criteria:

* HIV infection
* Chronic paraphimosis
* Genital ulcers
* Penile carcinoma
* Filariasis
* Xerotica obliterans
* Balanitis
* Glans-prepuce adhesions
* Frenular scar tissue
* Urethral anatomical abnormality such as hypospadias or epispadias

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Procedure Time | 21 days
  Primary outcomes of interest was procedure time. An assistant measured operative time using a stopwatch. For the SR group, timing began as the ring began to be fitted, and ceased when the foreskin had been excised. For the FG group, timing began at the first incision and ceased when the final suture was completed.
Major Complication | 21 days
  We considered a major complication as one requiring assessment by a clinician, including any of: a) SR slippage; b) infection requiring antibiotics, or c) any persistent complication on day 14.

SECONDARY OUTCOMES:
Pain | 21 days
  Pain scales were measured on post-op day 1, 3, 7, 14, and 21 using a visual analogue scale.
Time to resumption of normal activity | 21 days
  Self-reported time to resumption of normal activity (defined as attendance at university classes)
Patient Satisfaction | 21 days
  Patient satisfaction taken at conclusion of follow-up (rated as 'low', 'average', 'high' or "very high" and dichotomized as low/average or high/very high for analyses)
Time to complete healing | 21 days
  As measured by primary surgeon (study primary investigator) at follow-up visits. Missing outcome data for patients in the FG group who did not return were allocated as favourable for analysis of outcomes to bias estimates of a superiority of the SR towards the null. Thus, for patients in the FG group who did not return, we considered them to have high satisfaction and no major complications.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Kanyago, MD, Principal Investigator — Mbarara University of Scince and Technology
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

REFERENCES:
- [Background] Siegfried N, Muller M, Volmink J, Deeks J, Egger M, Low N, Weiss H, Walker S, Williamson P. Male circumcision for prevention of heterosexual acquisition of HIV in men. Cochrane Database Syst Rev. 2003;(3):CD003362. doi: 10.1002/14651858.CD003362. PMID 12917962
- [Background] Auvert B, Taljaard D, Lagarde E, Sobngwi-Tambekou J, Sitta R, Puren A. Randomized, controlled intervention trial of male circumcision for reduction of HIV infection risk: the ANRS 1265 Trial. PLoS Med. 2005 Nov;2(11):e298. doi: 10.1371/journal.pmed.0020298. Epub 2005 Oct 25. PMID 16231970
- [Background] Bailey RC, Moses S, Parker CB, Agot K, Maclean I, Krieger JN, Williams CF, Campbell RT, Ndinya-Achola JO. Male circumcision for HIV prevention in young men in Kisumu, Kenya: a randomised controlled trial. Lancet. 2007 Feb 24;369(9562):643-56. doi: 10.1016/S0140-6736(07)60312-2. PMID 17321310
- [Background] Gray RH, Kigozi G, Serwadda D, Makumbi F, Watya S, Nalugoda F, Kiwanuka N, Moulton LH, Chaudhary MA, Chen MZ, Sewankambo NK, Wabwire-Mangen F, Bacon MC, Williams CF, Opendi P, Reynolds SJ, Laeyendecker O, Quinn TC, Wawer MJ. Male circumcision for HIV prevention in men in Rakai, Uganda: a randomised trial. Lancet. 2007 Feb 24;369(9562):657-66. doi: 10.1016/S0140-6736(07)60313-4. PMID 17321311
- [Background] Barone MA, Ndede F, Li PS, Masson P, Awori Q, Okech J, Cherutich P, Muraguri N, Perchal P, Lee R, Kim HH, Goldstein M. The Shang Ring device for adult male circumcision: a proof of concept study in Kenya. J Acquir Immune Defic Syndr. 2011 May 1;57(1):e7-12. doi: 10.1097/QAI.0b013e3182158967. PMID 21346586